CLINICAL TRIAL: NCT04354480
Title: A Randomized, Double-blind, Placebo-controlled, Phase 1 Study to Evaluate the Safety, Reactogenicity and Immunogenicity of Single Vaccination of an Ad26.RSV.preF-based Regimen in Japanese Adults Aged 60 Years and Older
Brief Title: A Study to Evaluate the Single Vaccination of an Adenovirus Serotype 26 Pre-Fusion F (Ad26.preF) Based Respiratory Syncytial Virus (RSV) Vaccine in Japanese Adults Aged 60 Years and Older
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CR108768; VAC18193RSV1006 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — Respiratory Syncytial Virus Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- RSV Vaccine (Experimental): Participants will receive a single intramuscular (IM) injection of an adenovirus serotype 26 (Ad26)-based respiratory syncytial virus (RSV) vaccine at a single dose level on Day 1.
  Interventions: Biological: RSV Vaccine
- Placebo (Placebo Comparator): Participants will receive single IM injection in the deltoid muscle of matching placebo on Day 1.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: RSV Vaccine — Participants will receive single IM injection of Ad26.preF RSV based vaccine on Day 1.
  Arms: RSV Vaccine
Other: Placebo — Participants will receive a single IM injection of matching placebo on Day 1.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to assess the safety and reactogenicity of the Ad26.preF based RSV vaccine administered intramuscularly as a single injection versus placebo in Japanese adults aged greater than equal to 60 years.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be a Japanese participant whose parents and grandparents are Japanese as determined by the participant's verbal report
* Before randomization, a woman must be: postmenopausal (A postmenopausal state is defined as no menses for 12 months without an alternative medical cause); not intending to conceive by any methods
* A male participant must agree not to donate sperm for the purpose of reproduction for a minimum 28 days after receiving the dose of study vaccine
* In the investigator's clinical judgment, participant must be either in good or stable health. Participants may have underlying illnesses such as hypertension, type 2 diabetes mellitus, hyperlipoproteinemia, or hypothyroidism, as long as their symptoms/signs are medically controlled. If they are on medication for a condition, the medication dose must have been stable for at least 12 weeks preceding vaccination and expected to remain stable for the duration of the study. Participants will be included on the basis of physical examination, medical history, vital signs , and 12-lead electrocardiogram (ECG) performed at screening
* From the time of vaccination through 3 months, participant agrees not to donate blood
* Participant must be willing to provide verifiable identification, have means to be contacted and to contact the investigator during the study

Exclusion Criteria:

* Participant has a serious chronic disorder, including severe chronic obstructive pulmonary disease or clinically significant congestive heart failure, end stage renal disease with or without dialysis, clinically unstable cardiac disease, Alzheimer's disease, or has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (example, compromise well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Participant has history of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which is considered cured with minimal risk of recurrence)
* Participant has chronic active hepatitis B or hepatitis C infection, documented by hepatitis B surface antigen and hepatitis C antibody, respectively
* Participant has had major psychiatric illness and/or drug or alcohol abuse which in the investigator's opinion would compromise the participant's safety and/or compliance with the study procedures
* Participant has a history of chronic urticaria (recurrent hives), eczema and/or atopic dermatitis

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Solicited Local Adverse Events (AEs) After Vaccination | 7 days after vaccination (Day 1 to Day 8)
  Number of participants with solicited local AE's will be evaluated. Solicited local AEs (including erythema, swelling, and pain/tenderness at the study vaccine injection site) will be noted in the participant diary after 7 days of vaccination.
Number of Participants with Solicited Systemic Adverse Events (AEs) After Vaccination | 7 days after vaccination (Day 1 to Day 8)
  Number of participants with solicited systemic AEs will be evaluated. Solicited systemic AEs (fatigue, headache, myalgia, nausea and fever) will be noted in the participant diary after 7 days of vaccination.
Number of Participants with Unsolicited AEs | 28 days after vaccination (Day 1 to Day 29)
  Number of participants with unsolicited AEs will be evaluated. An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. Unsolicited AEs will include all AEs for which the participant is not specifically questioned in the participant diary.
Number of Participants with Serious Adverse Events (SAEs) | First vaccination (Day 1) to the end of the study (up to Day 183)
  Number of participants with SAEs will be evaluated. A SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life threatening experience, is a congenital anomaly/birth defect, is suspected transmission of any infectious agent via a medicinal product, is medically important, and may jeopardize participant or may require medical or surgical intervention to prevent one of the outcomes listed above.

SECONDARY OUTCOMES:
RSV Neutralization Assay | Day 1 (pre-vaccination), Days 14, 28, and 182 (post-vaccination)
  Analysis of neutralizing antibodies to RSV A strain will be performed.
RSV Fusion Protein (F-Protein) Binding Antibodies by Enzyme-linked Immunosorbent Assay (ELISA) | Day 1 (pre-vaccination), Days 14, 28, and 182 (post-vaccination)
  Antibodies binding to RSV F-protein in pre-fusion and post-fusion forms will be assessed by ELISA.
Interferon (IFN)-Gamma Enzyme-Linked Immunospot (ELISpot) Assay | Day 1 (pre-vaccination) and Day 29 (post-vaccination)
  RSV F-specific cellular immune responses elicited by the different vaccine regimens.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- Souseikai Hakata Clinic, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Eto T, Okubo Y, Momose A, Tamura H, Zheng R, Callendret B, Bastian AR, Comeaux CA. A Randomized, Double-Blind, Placebo-Controlled, Phase 1 Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of Single Vaccination of Ad26.RSV.preF-Based Regimen in Japanese Adults Aged 60 Years and Older. Influenza Other Respir Viruses. 2024 Jun;18(6):e13336. doi: 10.1111/irv.13336. PMID 38880785